CLINICAL TRIAL: NCT02797704
Title: The Effect of Subconjunctival Aflibercept on Regression of Corneal Neovascularization
Brief Title: Subconjunctival Aflibercept (EYLEA®) for the Treatment of Corneal Neovascularization
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: the treatment was found to be inefficient for all recruited patients
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0134-16-RMC
Record Dates: First submitted 2016-05-24; First posted 2016-06-13 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2016-05

CONDITIONS: Corneal Neovascularization
MeSH Terms: conditions — Corneal Neovascularization | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SC Aflibercept (Experimental): The patients will be treated with a single subconjunctival injection of 0.08 ml aflibercept (25 mg/ml) in a single quarter of the conjunctiva, near the limbus in a proximity to the area of pathological neovascularization
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Eylea (aflibercept) Injection is a prescription medicine administered by injection into the eye.
  Other Names: Eylea

SUMMARY:
The goal of this current study is to prospectively evaluate the influence of a single subconjunctival aflibercept injection on the regression of corneal neovascularization. Twenty patients with corneal neovascularization who are candidates for anti VEGF treatment (by the discretion of a corneal specialist) will be included in this study. The patients will be treated with a single subconjunctival injection of 0.08 ml aflibercept (25 mg/ml) in a single quarter of the conjunctiva, near the limbus in a proximity to the area of pathological neovascularization. Regression of neovascularization will be documented.

DETAILED DESCRIPTION:
An interruption of the equilibrium between proangiogenic and antiangiogenic factors in the usually nonvascularized cornea causes new corneal vessels to sprout, interfering with the corneal clarity that is essential for maintaining normal vision. Treating the neovascularized and often scarred cornea remains highly challenging because the loss of immunologic privilege in the avascular cornea makes it a poor candidate for corneal transplantation.

Vascular endothelial growth factor (VEGF) is a key cytokine in the development of both normal blood vessels and vessels in tumors and other tissues undergoing abnormal angiogenesis. In the cornea, VEGF is one of several known mediators of neovascularization. In recent years, anti-VEGF compounds have been extensively investigated for use in the prevention and treatment of neovascularization in many tissues, including the cornea. Experimental models and clinical studies have reported promising results for such anti-VEGF compounds as bevacizumab (Avastin®) and ranibizumab (Lucentis®). Aflibercept is a VEGF-Trap molecule. It has the highest affinity of all VEGF blockers studied to date. Aflibercept has been approved in the United States and Europe for the treatment of macular degeneration under the trade name Eylea® and the treatment of metastatic colorectal cancer under the trade name Zaltrap®. It has been found to offer a more prolonged and potentially more potent anti-VEGF effect in wet age-related macular degeneration than both bevacizumab and ranibizumab. Aflibercept's safety has been proven for this indication.

A preliminary study in a rat model recently conducted by our group demonstrated that subconjunctival (SC) injection and topical administration of aflibercept efficiently prevented corneal neovascularization compared to bevacizumab. The aim of this present study is to determine aflibercept's efficacy in the treatment of corneal neovascularization in humans.

Goal:

To prospectively evaluate the influence of a single subconjunctival aflibercept injection on the regression of corneal neovascularization.

Design and Clinical Follow-up:

A prospective study, including patients with various corneal pathologies complicated by corneal neovascularization.

Twenty patients with corneal neovascularization who are candidates for anti VEGF treatment (by the discretion of a corneal specialist) will be included in this study. The patients will be treated with a single subconjunctival injection of 0.08 ml aflibercept (25 mg/ml) in a single quarter of the conjunctiva, near the limbus in a proximity to the area of pathological neovascularization.

During follow-up period, previous medical and ophthalmic history will be documented. On the first visit, a thorough eye examination will be performed (including: Best Corrected Visual Acuity (BCVA), slit lamp examination of anterior segment including fluorescein staining of cornea for the assessment of epithelial integrity, intraocular pressure (IOP) measurements with Goldman tonometry, and a specular microscopy examination). Follow-up examinations will occur on days 7, 14, 30, 60, 90 following injection. Each follow-up meeting will include documentation of BCVA, IOP, a slit lamp exam and specular microscopy exam. Investigators will also perform anterior segment color photography before injection and at the last visit to document regression of neovascularization.

If no improvement or partial improvement is noted on the 30th day follow-up, the cornea specialist will consider a repeat subconjunctival aflibercept injection.

ELIGIBILITY:
Inclusion Criteria:

In this study, included will be patients with corneal neovascularization secondary to various pathologies, including: Pterygium, Corneal chemical burn, S/P corneal transplantation, Herpetic keratitis, atopic keratoconjunctivitis, Chronic retinal detachment, Uveitis, panus secondary to blepharitis, S/P corneal foreign body.

Exclusion Criteria:

1. Patients with a history of retinal vein/artery occlusion or diabetes, currently treated with anti-VEGF or with a history of such treatment 3 months prior to enrollment.
2. Prior treatment for corneal neovascularization with the injection of Avastin/Lucentis.
3. Patients under 18
4. Pregnant women
5. Contra indications for Eylea treatment, including intraocular or periocular infection/inflammation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Regression (change from baseline) of neovascularization clinically assessed by a corneal specialist | 3 months (90 days), with repeat assessment at different follow up times at 7,14,30,60 and 90 days.
  Regression of corneal neovascularization as the change from baseline will be assessed at all follow-up times on days 7,14,30,60,90 following injection by the corneal specialist, both by a clinical slit lamp exam to evaluate the area of neovascularization from the entire corneal area (which will be determined clinically by the ophthalmologist), and by performing anterior segment color photography before injection and at the last visit for comparison and documentation purposes.

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | 3 months
  BCVA will be assessed using a Snellen Chart at all follow-up meetings, and converted to logMAR for statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Irit Bahar, MD, Principal Investigator — Head of ophthalmology department
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Background] Azar DT. Corneal angiogenic privilege: angiogenic and antiangiogenic factors in corneal avascularity, vasculogenesis, and wound healing (an American Ophthalmological Society thesis). Trans Am Ophthalmol Soc. 2006;104:264-302. PMID 17471348
- [Background] Stevenson W, Cheng SF, Dastjerdi MH, Ferrari G, Dana R. Corneal neovascularization and the utility of topical VEGF inhibition: ranibizumab (Lucentis) vs bevacizumab (Avastin). Ocul Surf. 2012 Apr;10(2):67-83. doi: 10.1016/j.jtos.2012.01.005. Epub 2012 Jan 25. PMID 22482468
- [Background] Dastjerdi MH, Sadrai Z, Saban DR, Zhang Q, Dana R. Corneal penetration of topical and subconjunctival bevacizumab. Invest Ophthalmol Vis Sci. 2011 Nov 7;52(12):8718-23. doi: 10.1167/iovs.11-7871. PMID 22003112
- [Background] Chang JH, Garg NK, Lunde E, Han KY, Jain S, Azar DT. Corneal neovascularization: an anti-VEGF therapy review. Surv Ophthalmol. 2012 Sep;57(5):415-29. doi: 10.1016/j.survophthal.2012.01.007. PMID 22898649
- [Background] Chang JH, Gabison EE, Kato T, Azar DT. Corneal neovascularization. Curr Opin Ophthalmol. 2001 Aug;12(4):242-9. doi: 10.1097/00055735-200108000-00002. PMID 11507336
- [Background] Oliveira HB, Sakimoto T, Javier JA, Azar DT, Wiegand SJ, Jain S, Chang JH. VEGF Trap(R1R2) suppresses experimental corneal angiogenesis. Eur J Ophthalmol. 2010 Jan-Feb;20(1):48-54. doi: 10.1177/112067211002000106. PMID 19882518
- [Background] Rocher N, Behar-Cohen F, Pournaras JA, Naud MC, Jeanny JC, Jonet L, Bourges JL. Effects of rat anti-VEGF antibody in a rat model of corneal graft rejection by topical and subconjunctival routes. Mol Vis. 2011 Jan 11;17:104-12. PMID 21245949
- [Background] Semeraro F, Morescalchi F, Duse S, Parmeggiani F, Gambicorti E, Costagliola C. Aflibercept in wet AMD: specific role and optimal use. Drug Des Devel Ther. 2013 Aug 5;7:711-22. doi: 10.2147/DDDT.S40215. eCollection 2013. PMID 23990705
- [Result] Dratviman-Storobinsky O, Avraham-Lubin BCR, Hasanreisoglu M, Goldenberg-Cohen N. Effect of subconjuctival and intraocular bevacizumab injection on angiogenic gene expression levels in a mouse model of corneal neovascularization. Mol Vis. 2009 Nov 13;15:2326-38. PMID 19936307
- [Result] Avisar I, Weinberger D, Kremer I. Effect of subconjunctival and intraocular bevacizumab injections on corneal neovascularization in a mouse model. Curr Eye Res. 2010 Feb;35(2):108-15. doi: 10.3109/02713680903429007. PMID 20136420
- [Result] Habot-Wilner Z, Barequet IS, Ivanir Y, Moisseiev J, Rosner M. The inhibitory effect of different concentrations of topical bevacizumab on corneal neovascularization. Acta Ophthalmol. 2010 Dec;88(8):862-7. doi: 10.1111/j.1755-3768.2009.01571.x. PMID 19549103
- [Result] Park YR, Chung SK. Inhibitory Effect of Topical Aflibercept on Corneal Neovascularization in Rabbits. Cornea. 2015 Oct;34(10):1303-7. doi: 10.1097/ICO.0000000000000507. PMID 26114826
- [Result] Sella R, Gal-Or O, Livny E, Dachbash M, Nisgav Y, Weinberger D, Livnat T, Bahar I. Efficacy of topical aflibercept versus topical bevacizumab for the prevention of corneal neovascularization in a rat model. Exp Eye Res. 2016 May;146:224-232. doi: 10.1016/j.exer.2016.03.021. Epub 2016 Mar 26. PMID 27020759
- [Result] Gal-Or O, Livny E, Sella R, Nisgav Y, Weinberger D, Livnat T, Bahar I. Efficacy of Subconjunctival Aflibercept Versus Bevacizumab for Prevention of Corneal Neovascularization in a Rat Model. Cornea. 2016 Jul;35(7):991-6. doi: 10.1097/ICO.0000000000000849. PMID 27124775